CLINICAL TRIAL: NCT00305890
Title: Duke University Pain Prevention: Weight Management and Coping Skills Training For Patients With Osteoarthritis of the Knee
Brief Title: Weight Management and Coping Skills Training For Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008156; P01AR050245 (NIH); NIAMS-4927; 1P01AR050245-03 (NIH)
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2013-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants will partake in a lifestyle behavioral weight management program for 24 weeks.
  Interventions: Behavioral: Lifestyle Behavioral Weight Management Program
- 2 (Experimental): Participants will partake in pain-coping skills training for 24 weeks.
  Interventions: Behavioral: Pain-Coping Skills Training
- 3 (Experimental): Participants will partake in lifestyle behavioral weight management program plus pain-coping skills training for 24 weeks.
  Interventions: Behavioral: Lifestyle Behavioral Weight Management Program; Behavioral: Pain-Coping Skills Training
- 4 (Active Comparator): Participants will receive standard care for 24 weeks.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Lifestyle Behavioral Weight Management Program — The lifestyle behavioral weight management program will focus on lifestyle, exercise, attitudes, relationships, and nutrition. Participants will attend 12 weekly group sessions, followed by 6 every-other-week group sessions.
  Arms: 1; 3
Behavioral: Pain-Coping Skills Training — The pain-coping skills training will focus on minimizing maladaptive over-reactions and enhancing adaptive strategies to control and decrease pain. Participants will attend 12 weekly group sessions, followed by 6 every-other-week group sessions.
  Arms: 2; 3
Other: Standard Care — Standard care will include routine medical care.
  Arms: 4

SUMMARY:
Osteoarthritis (OA) occurs when the cartilage between two bones becomes worn down, and the bones begin to rub against each other in the joint. This often leads to pain, swelling, decreased joint motion, and the formation of bone spurs (tiny growths of new bone). Being overweight increases the risk of developing OA and fastens disease progression. This study will evaluate two different programs, lifestyle behavioral weight management and pain-coping skills training, in reducing the effects of knee OA in obese individuals.

DETAILED DESCRIPTION:
Osteoarthritis is a chronic, degenerative joint disorder that does not have a cure. While OA can occur at almost any joint, it most commonly occurs in the knee. Obesity is a significant risk factor for the development of knee OA and is associated with faster disease progression. Biomechanical inflammation and cognitive behavioral changes related to obesity can exacerbate OA pain and disability. The purpose of this study is to develop more effective ways to treat individuals with knee OA. Specifically, the study will compare the effectiveness of a lifestyle behavioral weight management program, pain-coping skills training, and standard care in improving OA symptoms and day-to-day function in obese individuals with OA in one or both knees.

The study treatment groups will meet for a total of 6 months. Participants will be randomly assigned to one of four conditions: 1) lifestyle behavioral weight management program, 2) pain-coping skills training, 3) lifestyle behavioral weight management program plus pain-coping skills training, or 4) standard care. The lifestyle behavioral weight management program will focus on lifestyle, exercise, attitudes, relationships, and nutrition. The pain-coping skills training will focus on minimizing maladaptive over-reactions and enhancing adaptive strategies to control and decrease pain. Standard care will include routine medical care.

Participants in the first three conditions will attend 12 weekly group sessions, followed by 6 every-other-week group sessions. After completing treatment, participants will receive monthly follow-up telephone calls to facilitate the post-treatment transition. There will be a total of four evaluations during this study: immediately prior to treatment, immediately after treatment, and 6 and 12 months following the end of treatment. During each evaluation, blood and urine will be collected to analyze disease biomarkers. An exercise treadmill test and height, weight, and body mass index measures will be used to assess aerobic fitness. Lower extremity function will be measured with the "Up and Go" performance test. Participants will also be videotaped while walking to evaluate gait and will be asked to fill out a series of questionnaires. Medication use will be reviewed during an interview. During the first evaluation, x-rays will be taken to measure disease activity.

Participants completing the study intervention and all four follow-up evaluations will be eligible to join the second part of the study examining the relationship between food intake, mood, activity level, and pain. Participants will complete a series of questionnaires at baseline and 2-day diaries in which they rate mood, pain, and activity level and they record food intake triggered at random times throughout the day. A follow-up visit to complete additional questionnaires will be conducted 6 months later. Blood samples will also be collected for future analysis of genetic markers of pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Meets the American College of Rheumatology criteria for OA
* Radiographic evidence of OA affecting one or both knees
* Complaints of chronic knee pain (pain on most days for at least 6 months prior to study entry)
* No other major weight-bearing joint affected by OA

Exclusion Criteria:

* Any significant medical condition or disease that would make study participation unsafe or increase the risk of a significant adverse experience during the course of the study (e.g., myocardial infarction in the 6 months prior to study entry)
* Currently involved in a regular exercise program
* An abnormal cardiac response to exercise, such as exercise-induced BT or an abnormal blood pressure response
* A body mass index (BMI) greater than 42
* A non-OA inflammatory arthropathy
* Currently using oral corticosteroids on a regular basis
* Anticipate to have a knee surgery in the next 18 months (or before the anticipated date of their study completion)
* Knee surgery (arthroscopic or knee replacement) within a year of enrollment
* Intraarticular steroid or hyaluronan knee injections in one of both knees within 3 months of enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2004-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Psychological impairment | Measured immediately, 6 months, and 12 months following treatment: pain
Physical disability | Measured immediately, 6 months, and 12 months following treatment: pain
Joint stiffness | Measured immediately, 6 months, and 12 months following treatment: pain
Activity level | Measured immediately, 6 months, and 12 months following treatment: pain
Physical activities | Measured immediately, 6 months, and 12 months following treatment: pain

SECONDARY OUTCOMES:
Physiological measures of disease activity | Measured immediately, 6 months, and 12 months following treatment: pain
Gait measures | Measured immediately, 6 months, and 12 months following treatment: pain

CONTACTS AND LOCATIONS:
Overall Officials: Francis Keefe, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Morreene Rd. Clinic, Durham, North Carolina, United States

REFERENCES:
- [Derived] Huebner JL, Landerman LR, Somers TJ, Keefe FJ, Guilak F, Blumenthal JA, Caldwell DS, Kraus VB. Exploratory secondary analyses of a cognitive-behavioral intervention for knee osteoarthritis demonstrate reduction in biomarkers of adipocyte inflammation. Osteoarthritis Cartilage. 2016 Sep;24(9):1528-34. doi: 10.1016/j.joca.2016.04.002. Epub 2016 Apr 16. PMID 27090577